CLINICAL TRIAL: NCT06987084
Title: A Novel Treatment for Recurrent Kidney Stones
Brief Title: Bryophyllum Pinnatum Tea as a Novel Treatment for Recurrent Kidney Stone Formers
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indra Gupta (Other)
Responsible Party: Sponsor-Investigator, Indra Gupta, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-8588
Record Dates: First submitted 2025-05-06; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Kidney Calculi; Calcium Oxalate Kidney Stones; Calcium Phosphate Kidney Stones
Keywords: Kidney stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Each participant will be assigned to one of the following groups:
  Group 1: Drink wheat-bran tea (placebo) first then, B. pinnatum tea (treatment).
  Group 2: Drink B. pinnatum tea first (treatment), then wheat-bran tea (placebo).
  The placebo and the treatment are sweetened with 1/2 teaspoon of sugar.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the B. pinnatum tea and the placebo tea will be provided in identical dark thermoses with a lid. The placebo wheat-bran tea tastes and looks identical to the treatment, B. pinnatum tea.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- B. pinnatum tea - First (Experimental): Participants in this arm will receive 250 mL of sweetened B. pinnatum tea on day 1 and then on day 2, they will submit urine and blood for analysis for biochemistry. On day 10, participants will receive 250 mL of sweetened placebo tea. On day 11, they will again submit a 24-hour urine collection and a blood sample for analysis.
  Interventions: Combination Product: Bryophyllum pinnatum tea; Combination Product: Placebo tea
- Placebo - First (Experimental): Participants in this arm will receive 250 mL of sweetened placebo tea on day 1 and then on day 2, they will submit urine and blood for analysis for biochemistry. On day 10, participants will receive 250 mL of sweetened B. pinnatum tea. On day 11, they will again submit a 24-hour urine collection and a blood sample for analysis.
  Interventions: Combination Product: Bryophyllum pinnatum tea; Combination Product: Placebo tea

INTERVENTIONS:
Combination Product: Bryophyllum pinnatum tea — 24 g of B. pinnatum leaves boiled in 250 mL of water for 61 minutes sweetened with 1/2 teaspoon of sugar
Combination Product: Placebo tea — 250 mL of water boiled with 3 g of wheat-bran for 5 minutes sweetened with 1/2 teaspoon of sugar

SUMMARY:
The aim of this randomized placebo-controlled double-blind crossover clinical trial is to test the ability of a traditional tea made from the leaf of the Bryophyllum pinnatum (B. pinnatum) plant in decreasing urinary calcium content in patients with recurrent calcium-based kidney stones.

DETAILED DESCRIPTION:
Background and Rationale:

Kidney stones are hard deposits that consist of calcium complexed with phosphate or oxalate, thus, high urinary calcium content is a major risk factor. The precipitation of calcium can arise from various mechanisms including the aggregation of urinary calcium crystals from impaired transport along the nephron, reduced urinary inhibitors (e.g. citrate), and increased oxidative stress and inflammation. Large stones can block the drainage system of the kidney, causing acute severe pain and inflammation. Recurrent kidney stones can lead to sustained inflammation resulting in a progressive loss of renal function. As the global incidence and economic burden continues to rise there is a undisputed medical need to find preventative measures.

Thiazide diuretics have been fundamental in pharmacological recurrence prevention for the past 60 years. The recent NOSTONE trial (NCT03057431) revealed that the most widely prescribed and best studied thiazide, hydrochlorothiazide, did not reduce the incidence of stone recurrence. There remain significant barriers to kidney stone treatment including high treatment costs, side effects, and the difficulty in achieving long-term dietary and lifestyle changes. Therefore, many patients risk recurrent episodes. New innovative approaches are needed to prevent kidney stone formation.

The leaves of Bryophyllum pinnatum are used to treat a variety of ailments, including the prevention and treatment of kidney stones in various formulations. In a rat kidney stone model, aqueous, alcoholic, and non-alcoholic extracts of B. pinnatum leaves prevented the formation and reduced the size of kidney stones. In an uncontrolled trial, patients with renal stones treated with B. pinnatum juice either passed their stones or showed a reduction in the size of their stones. Despite its established use in other countries, B. pinnatum tea has not undergone rigorous scientific or clinical evaluation. Our lab characterized and standardized the formulation of the tea which revealed anti-urolithiatic activity along with antioxidant and anti-inflammatory properties. A combination of these effects may be what is beneficial in the prevention of recurrent kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age at time of study enrollment
* 1 calcium-based stone event within a 3-year interval and/or hypercalciuria on a 24h urine collection (>5 mmol/day)
* They had an ultrasound or CT imaging within the previous 6 months which showed no evidence of current obstructive kidney stone
* Adhering to the stone prevention diet (high water/low salt/low protein intake) for at least one month prior to enrollment in study but not taking any stone-preventing medications
* Agrees to maintain current lifestyle habits and avoid taking new supplements during the study period

Exclusion Criteria:

* Patients with secondary causes for calcium stone formation (primary hyperparathyroidism, inflammatory bowel disease, hyperuricosuria, and cancer)
* Patients who are pregnant or nursing or who are trying to become pregnant
* Currently consuming B. pinnatum or any natural health product containing polyphenols
* A known intolerance or allergy to the plant B. pinnatum
* Currently taking stone-preventing medication
* Gluten intolerance or allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in 24-hour urine calcium excretion | 24 hours after ingestion (day 2 and day 11)
  After ingestion of the placebo and treatment, participants will begin a 24 hour urine collection. Urinary calcium levels will be reported as mmol/day.

SECONDARY OUTCOMES:
Adverse effects | 24 hours after ingestion (day 2 and day 11)
  Partipants will be asked if they experience any adverse effects immediately after and 24 hours after ingestion.
Increase in 24-hour urine citrate excretion | 24 hours after ingestion (day 2 and day 11)
  After ingestion of the placebo and treatment, participants will begin a 24 hour urine collection. Urinary citrate levels will be reported as mmol/day.

CONTACTS AND LOCATIONS:
Overall Officials: Indra Gupta, MD, Principal Investigator — Research Institute at the McGill University Health Centre
Locations (1):
- McGill University Health Centre (Glen Site), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All anonymized patient data that underlies results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available 6 months after publication.
Access Criteria: All data will be anonymized for publication. Only the study investigators will have access to individual patient data.

REFERENCES:
- [Background] Chik C, Larroque AL, Zhuang Y, Feinstein S, Smith DL, Andonian S, Ryan AK, Jean-Claude B, Gupta IR. A Nuclear Magnetic Resonance (NMR)- and Mass Spectrometry (MS)-Based Saturation Kinetics Model of a Bryophyllum pinnatum Decoction as a Treatment for Kidney Stones. Int J Mol Sci. 2024 May 12;25(10):5280. doi: 10.3390/ijms25105280. PMID 38791318